CLINICAL TRIAL: NCT04755998
Title: Evaluating the Effect of the Use of Virtual Reality Headset in School Vaccinations on Children's Fear and Anxiety Levels
Brief Title: Evaluating the Effect of the Use of Virtual Reality Headset in School Vaccinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, İlknur KAHRİMAN, Assoc. Prof., Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: İlknur KAHRİMAN
Record Dates: First submitted 2021-02-13; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Anxiety and Fear
Keywords: Anxiety, Child, Fear, Vaccine, Virtual reality headset
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The Experimental Group watched cartoons with virtual reality glasses during vaccination applications.
  Interventions: Other: Use of virtual reality glasses during vaccination applications in children
- Control Group (No Intervention): Pre-test and post-tests were applied to the non-intervention group

INTERVENTIONS:
Other: Use of virtual reality glasses during vaccination applications in children — To the experimental group:
  Before the vaccine administration;
  * Children's Fear Scale, and Children's Anxiety Scale-State Scale was applied to the student.
  * Cartoons and virtual reality glasses that the student wanted to watch were prepared.
  * While the nurse was preparing the vaccines, the student was put on virtual reality glasses and the distance settings of the lenses were adjusted and the cartoons he chose to watch during the vaccination applications started to be shown. Since virtual reality glasses can cause anxiety attacks manifested by nausea in some children, this was also tested beforehand. It took about two minutes to administer the vaccine and watch cartoons.
  Those applied after the vaccine administration;
  - Children's Fear Scale, and Children's Anxiety Scale-State Scale was applied to the student.
  Arms: Experimental Group

SUMMARY:
This study was conducted with a randomized controlled experimental design to determine the effect of virtual reality headset on children's fear and anxiety during vaccinations.

Research Hypotheses:

Hypothesis 0a (H0a): There is no difference in fear scores between the experimental group in which virtual reality glasses were used during vaccination administration and the control group.

Hypothesis 1a (H1a): There is a difference in fear scores between the experimental group in which virtual reality glasses were used during vaccination administration and the control group.

Hypothesis 0b (H0b): There is no difference in anxiety scores between the experimental group in which virtual reality glasses were used during vaccination administration and the control group.

Hypothesis 1b (H1b): There is a difference in anxiety scores experienced between the experimental group in which virtual reality glasses were used during vaccination administration and the control group.

DETAILED DESCRIPTION:
Interventions made for protecting health or curing diseases, significantly affect children's psychological state and social adaptation. Being one of these interventions, vaccination may cause fear and anxiety in children. This fear and anxiety may affect children's future treatment and care experiences and result in fright and avoidance in them. Thus, it is important to try and reduce biological stress and to cope with psychosocial stress. One of the methods which can be used for this purpose is virtual reality headset used as a distraction method. This study was conducted with a randomized controlled experimental design to determine the effect of virtual reality headset on children's fear and anxiety during vaccinations. The population of the study consisted of first grade students attending primary schools in the city center of Ordu. The study was completed with 84 students in the experimental group and 85 students in the control group. With the sample number obtained as a result of the study, the test power was found to be 89.8% when the alpha error was 0.05 and the effect size was kept at 0.5. The data were collected using the Child and Parent Introductory Information Form, Children's Fear Scale, and Children's Anxiety Scale-State Scale.

ELIGIBILITY:
Inclusion Criteria:

* Parental consent
* Student's willingness to participate in the research
* The student does not have a mental or neurological disability
* Not being able to communicate
* The student does not have a chronic illness
* The student does not have an illness that causes acute or chronic pain
* The student has not used any analgesic medication in the last 24 hours.

Exclusion Criteria:

* Lack of parental consent
* Student's unwillingness to participate in the research
* The student has a mental or neurological disability
* The student has a communication disability
* The student has a chronic illness
* The student has an illness that causes acute or chronic pain
* The student's use of medication that will have an analgesic effect in the last 24 hours.

Ages: 72 Months to 84 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 169 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The Child Fear Scale | with an average interval of three to five minutes
  This scale is a one-item self-report measure for measuring pain-related fear in children. This one-item scale consists of five sex-neutral faces. It ranges from a no fear (neutral) face on the far left to a face showing extreme fear on the far right. It can be used for children aged 5-10 years.
The Children's Anxiety Scale-State Scale | with an average interval of three to five minutes
  It assesses children's anxiety in clinical settings and uses before medical procedures. The Children's Anxiety Scale-State Scale is drawn like a thermometer with a bulb at the bottom, also includes horizontal lines at intervals going up to the top. Children are asked to mark how he/she feel "right now" to measure state anxiety. Scores range from 0 to 10. It validated at children aged 4-10 years during an intravenous procedure.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur KAHRİMAN, Assoc. Prof., Study Director — Karadeniz Technical University; Zila Ö KIRBAŞ, Master, Principal Investigator — Karadeniz Technical University
Locations (1):
- DIRECTORATE OF PROVINCIAL EDUCATION, and PROVINCIAL HEALTH DIRECTORATE, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: CSR
Time Frame: 12 months after publication
Access Criteria: Relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.